CLINICAL TRIAL: NCT04451993
Title: Are the Sleep Quality and Physical Activity Levels of Osas Patients Differently From Healthy People During the COVID-19 Pandemic:a Prospective, Descriptive Study
Brief Title: Physical Activity Level in Patients With OSAS During Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, NUREL ERTURK, Phd student, Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital
Other Study IDs: GO 20/540
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea-hypopnea Syndrome
Keywords: physical activity; COVID-19; sleep quality
MeSH Terms: conditions — Motor Activity; COVID-19; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSAS PATIENTS: mild, moderate and severe OSAS patients
- HEALTHY INDIVIDUALS: healthy individuals without chronic disease

SUMMARY:
As long as the people stay at home because of the Covid 19 outbreak, the investigators assume that the sleep quality of OUAS patients, like everyone else, and the sleep quality of COVID-19 outbreak are reduced due to anxiety and anxiety in people. In addition, we assume that sleep quality and physical activity level are related to health literacy level and fear of movement (kinesiophobia). In this study; the investigators aimed to determine how patients are affected by this process by evaluating sleep quality, physical activity, fear of movement and health literacy in OSAS patients during our stay in the COVID-19 outbreak.

DETAILED DESCRIPTION:
Research Ahi Evren Chest Cardiovascular Surgery Training Research Hospital will be performed in patients between the ages of 18-70 years, diagnosed with OSAS in the sleep laboratory. Sleep quality, physical activity, fear of movement and health literacy will be evaluated in OSAS patients. Evaluations will be made by phone In order for the study to be strong, it will be tried to reach the maximum patient that can be taken between June 2020 and October 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Having been diagnosed with OSAS and disease severity determined,
2. Being between the age of 19-70,
3. Body mass index <40 kg / m2
4. Volunteering to participate in the research,
5. Not having a mental problem that will hinder the cooperation.

Exclusion Criteria:

1. To have advanced orthopedic, neurological and cardiovascular disease,
2. Having a cognitive problem,

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy individuals between 18-70 years old, who are diagnosed with OSAS in the sleep lab at the Ahi Evren Chest, Heart and Vascular Surgery Training and Research Hospital, and whose local language is Turkish will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 1 day
  International Physical Activity Questionnaire/ In activity-specific scoring, walking under the heading of the fields is calculated by the sum of the moderate intensity activity and intensive activity in itself.
  From these calculations, a score is obtained in MET-minutes. There are 3 categories of physical activity level classification. Physical activity levels are classified as physically inactive (inactive), low level of physical activity (minimally active) and sufficient level of physical activity (very active)
Sleep Quality | 1 day
  The Pittsburgh Sleep Quality Index

SECONDARY OUTCOMES:
Daytime Sleepiness | 1 day
  In order to measure the general sleepiness of people during the day, it was evaluated with a standard questionnaire, which is defined as Epworth sleepiness scale (EUS) and consists of 8 questions. The answers for each question are scored between 0 and 3 and the total score is obtained. The score obtained above 10 in EUS has high sensitivity and specificity for daytime sleepiness.
Fear of movement | 1 day
  Tampa Kinesiophobia Scale (TKS)The person gets a total score between 17-68. The high score on the scale indicates that kinesiophobia is also high
Health literacy | 1 day
  Translated into Turkish TURKEY health literacy SCALE-32 (Tsoy-32) will be used. It was used to evaluate the literacy rates of individuals over the age of 15.
  0 indicates the lowest health literacy and 50 indicates the highest health literacy.

OTHER OUTCOMES:
Circadian rhythm evaluation | 1 day
  In the human circadian rhythm, the Morning Morning-Evening Survey (SAA) form was used, which determined morning and evening types.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Adem Celik, MD, Study Chair — Ahi Evren Chest, Heart and Vascular Surgery Training and Research Hospital
Locations (1):
- Trabzon Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No